CLINICAL TRIAL: NCT01330264
Title: Study of ICP Monitoring in Critically Ill
Brief Title: Study of Intracranial Pressure (ICP) Monitoring in Critically Ill
Acronym: SIM City
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00016075
Record Dates: First submitted 2011-04-05; First posted 2011-04-06 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Intracranial Pressure
Keywords: Intracranial Pressure (ICP) Monitoring; Admission to Intensive Care Unit (ICU)

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dyad

SUMMARY:
The SIM City study seeks to explore for the variance in practice that is associated with nursing and medical care of patients with brain pressure (ICP) monitors. The underlying hypothesis is that there is not a consistent pattern of care throughout the U.S., rather, there is a wide range of practice patterns that are used to monitor and treat ICP.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age or older)
* Admitted to an Intensive Care Unit (ICU)

Exclusion Criteria:

* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU that are receiving Intracranial Pressure (ICP) monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DaiWai M Olson, PhD RN CCRN, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States